CLINICAL TRIAL: NCT03704558
Title: Preoperative Radiographic Evaluation of Medial Tibiofemoral Knee Osteoarthritis: Reproducibility, Reliability and Correlation With Ligament Injury
Brief Title: Preoperative Radiographic Evaluation of Medial Tibiofemoral Knee Osteoarthritis
Acronym: RX-FTI
Status: Withdrawn | Type: Observational
Why Stopped: The project leader has left the institution
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC18_3012_RX-FTI
Record Dates: First submitted 2018-10-10; First posted 2018-10-15 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Arthritis Knee

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational study.

DETAILED DESCRIPTION:
In advanced stage osteoarthritis or osteonecrosis of the articular bearing surfaces of the knee, the surgical therapeutic solutions consist of a replacement of the articular surfaces by prosthetic implants. Depending on whether these implants replace all or part of the articular surfaces they are called "total" or "uni compartmental" knee prosthesis.

The uni-compartmental medial prosthesis replaces only the medial tibiofemoral compartment of the knee and is therefore intended for patients with cartilaginous wear isolated from this compartment.

The uni-compartmental medial prosthesis has advantages over the total knee arthroplasty of being more economical in articular tissues of the knee, having better functional results and lower complication rates. Although this is debated, the survival rate of uni-compartmental prostheses in the international registers is lower than that of total knee prostheses.

One of the most common early failure factors of uni-compartmental prostheses is the absence of a functional anterior cruciate ligament. Other factors have also been identified and are sometimes highly debated such as the Kozinn and Scott criteria. The group of designers of the unicompartmental Oxford Uni compartmental prosthesis Knee Arthroplasty (OUKA) (Zimmer Biomet, Warsaw) proposed and validated expanded criteria. These criteria, exclusively radiographic, are grouped in a document called "decision aid" to check the functional status of the collateral ligaments medial and anterior cross, other compartments of the knee (lateral femoro-tibial and femoro-patellar).

In decision aid, the functional status of the anterior cruciate ligament is judged on the knee radiograph by the location of the osteoarthritic cup. If it is present and functional, the cartilaginous wear is anterior with a respect of the posterior portion of the tibial plateau.

After regular use of the French version of the decision aid, the assessment of the location of osteoarthritis seems subjective to us however it is essential to validate the indication of a uni-compartmental prosthesis. In case of poor evaluation, the risk is the intraoperative discovery of the actual status of the anterior cruciate ligament that may result in a change of indication and the installation of a total knee prosthesis. The investigators have not found in the literature, studies evaluating the reliability and reproducibility of the lateral radiograph to judge the functional status of the anterior cruciate ligament.

The hypothesis is that the lateral radiograph is unreliable and reproducible to judge the functional status of the anterior cruciate ligament in a population of patients with medial femoro-tibial knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or over;
* presenting with medial femoral tibial osteoarthritis;
* Indication of a TKA or a medial PUC of first intention;
* Validation of the surgical indication at orthopedic surgery staff;
* Not having expressed his opposition to participate in the study.

Exclusion Criteria:

* Major person subject to legal protection (safeguard of justice, guardianship, guardianship);
* Person deprived of liberty;
* Pregnant or nursing woman.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient who received a uni-compartmental prosthesis or a total knee replacement over a period of 6 months at the Rennes University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Correlation | Baseline
  Correlation rate between compliance with the posterior third of the radiologically assessed tibial plateau and the functional status of the anterior cruciate ligament

SECONDARY OUTCOMES:
Reproducibility | Baseline
  Inter and intra-observer reproducibility of the preoperative radiological analysis: size of the wear cup, distance posterior edge of the tray - cup, respect of the posterior third and functional status of the anterior cruciate ligament
Reliability | Baseline
  Reliability of profile radio: correlation rate between radiological and intraoperative data

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Gicquel, Principal Investigator — Rennes University Hospital